CLINICAL TRIAL: NCT05221801
Title: Trunk Inclination Angle on Swallowing/Respiratory Function and the Development of Smart Positioning-angle Adjustment Device
Brief Title: Trunk Inclination on Respiratory-swallowing Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 201600752A3
Record Dates: First submitted 2022-01-11; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2017-01

CONDITIONS: Disabling Disease
Keywords: positioning; swallowing; respiration; sensors; disability; assistive device
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: The measurement would be done in 4 seat inclination angles (5, 15, 30, 45) and for 3 different food types for each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- angle 5 + 1ml water (Active Comparator): The measurement would be done in seat inclination angles of 5 degrees with 1 ml water intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 5 + 5 ml water (Active Comparator): The measurement would be done in seat inclination angles of 5 degrees with 5 ml water intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 5 + 5 ml pudding (Active Comparator): The measurement would be done in seat inclination angles of 5 degrees with 5 ml pudding intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 15 + 1ml water (Active Comparator): The measurement would be done in seat inclination angles of 15 degrees with 1 ml water intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 15 + 5 ml water (Active Comparator): The measurement would be done in seat inclination angles of 15 degrees with 5 ml water intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 15 + 5 ml pudding (Active Comparator): The measurement would be done in seat inclination angles of 15 degrees with 5 ml pudding intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 30 + 1ml water (Active Comparator): The measurement would be done in seat inclination angles of 30 degrees with 1 ml water intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 30 + 5 ml water (Active Comparator): The measurement would be done in seat inclination angles of 30 degrees with 5 ml water intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 30 + 5 ml pudding (Active Comparator): The measurement would be done in seat inclination angles of 30 degrees with 5 ml pudding intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 45 + 1ml water (Active Comparator): The measurement would be done in seat inclination angles of 45 degrees with 1 ml water intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 45 + 5 ml water (Active Comparator): The measurement would be done in seat inclination angles of 45 degrees with 5 ml water intake.
  Interventions: Behavioral: angle of inclination; Other: food type
- angle 45 + 5 ml pudding (Active Comparator): The measurement would be done in seat inclination angles of 45 degrees with 5 ml pudding intake.
  Interventions: Behavioral: angle of inclination; Other: food type

INTERVENTIONS:
Behavioral: angle of inclination — The measurement would be done in seat inclination angles of 5,15,30,45 degrees.
Other: food type — the swallowing was tested with 3 food types

SUMMARY:
Most caregivers do not know the influence of improper positioning therefore subjects suffer from possible choking risks. The aims of this study were to investigate the timing and coordination of swallowing and respiration in 4 different seat inclination angles, with liquid and bolus. A self-developed wearable device to measure the submandibular muscle surface EMG, the movement of thyroid cartilage and respiratory status of nasal cavity. This program could auto-analysis the onset and offset of duration, and the excursion and strength of thyroid cartilage will be calculated when it was moving, coordination between breathing and swallowing was also included. The results of this study would serve as the clinical guidelines for proper feeding positions for different populations and for different food contents.

DETAILED DESCRIPTION:
Swallowing is not only an important function for life maintenance, but also for quality of life improvement. Statistics revealed that subjects with intellectual disability or multiple disabilities have problems in controlling muscle tone and maintaining posture. In such circumstances, these subjects experience problems during feeding or eating. The adjustment of seat inclination would help in feeding/eating process. However, the proper inclination angle should be evaluated by medical professionals, however, most caregivers do not know the influence of improper positioning therefore subjects suffer from possible choking risks. The aims of this study were to investigate the timing and coordination of swallowing and respiration in 4 different seat inclination angles, with liquid and bolus. In the first stage, the investigators intend to use a self-developed wearable device to measure the submandibular muscle surface EMG, the movement of thyroid cartilage and respiratory status of nasal cavity. This particular program could auto-analysis the onset and offset of duration, and the excursion and strength of thyroid cartilage will be calculated when it was moving, coordination between breathing and swallowing was also included. The measurement would be done in four seat inclination angles (5, 15, 30, 45) for each subject. The data collected between different conditions would be compared, and suggestions of ideal angles during swallowing would be made. The second stage is the design and development of a feedback-controlled seat angle adjustment device, based on the data collected. The results of this study would serve as the clinical guidelines for proper feeding positions for different populations and for different food contents. The ergonomic data would also provide references for assistive technology professionals and practitioners in device design and development.

ELIGIBILITY:
Inclusion Criteria:

Typical-developed:

1. ages ranged from 20 to 60 years old,

People with disabilities:

1. ages ranged from 20 to 60 years old,
2. usually a need for supplementary feeding.

Exclusion criteria:

* Excluded conditions are cases of intubation and feeding, severely mentally retarded or autistic cases that cannot express comfort, cases of frequent choking, and those who have been treated with a throat tube and have a narrow throat.
* Exclude subjects who have undergone throat or nasal cavity surgery or have abnormalities in these two parts

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Electromyography | 5 seconds before the beginning of the swallow to 5 seconds after the end of the swallow.
  Two electrodes were attached to the submandibular muscle to register the electric potential generated by the muscles.
thyroid cartilage excursion | 5 seconds before the beginning of the swallow to 5 seconds after the end of the swallow.
  A force-sensing resistor (FSR) was fixed over the larynx at the thyroid cartilage position with an elastic belt to detect the cartilage excursion.
nasal airflow | 5 seconds before the beginning of the swallow to 5 seconds after the end of the swallow.
  A nasal airflow cannula was placed in front of the nasal cavity and was connected to a pressure transducer (Pro-Tech Services, Murrysville, PA, USA) to detect exhalation and inhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Yi K Cheng, PhD, Principal Investigator — Chang Gung University, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan